CLINICAL TRIAL: NCT05462444
Title: The Research and Development of the Personalized Balanced Nutrition Concept in Kindergartens Through an IT Platform
Brief Title: Development of Personalized Balanced Nutrition Concept Through an IT Platform
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital Srebrnjak (Other)
Collaborators: IN2 Ltd. (Unknown)
Responsible Party: Principal Investigator, Mirjana Turkalj, MD, Professor, MD, PhD, Children's Hospital Srebrnjak
Other Study IDs: KK.01.1.1.07.0074
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Child Allergy; Allergic Reaction
Keywords: Allergy; Perosnalized nutrition; Obesity
MeSH Terms: conditions — Hypersensitivity; Obesity | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children with food allergy
  Interventions: Other: Skin prick test
- Children with food intolerance
  Interventions: Other: Skin prick test
- Children with other allergies (reference group)
  Interventions: Other: Skin prick test

INTERVENTIONS:
Other: Skin prick test — Skin prick test with a standard pallete of inhalational and nutritional allergens

SUMMARY:
By achieving effective cooperation between the Children's Hospital Srebrnjak (CHS), the Reference center for clinical allergology in children of the ministry of health, and IN2 Ltd., part of Constellation Software Inc., it is planned to develop an IT platform for the introduction of personalized balanced nutrition in kindergartens. The collected data which include the screening of the population, anthropometrical measurements, physical activity status, and medical examination, will be used to create a Registry of Allergies. Through the implementation of research activities, it is expected to develop an IT platform for personalized balanced nutrition of preschool children, which consists of a developed information system for continuous monitoring using a website and/or a mobile application.

DETAILED DESCRIPTION:
This study will involve kindergarten children (aged 1-6 years). The research takes place in six different phases: 1) development of the information system and data integration, 2) classification of target groups of kindergarten children according to nutritional status, 3) anthropometric monitoring of the development of kindergarten children, 4) establishment of an electronic register of allergies, 5) implementation of an information platform in kindergartens, and 6) assessment of the validity of platform. The research will include a minimum of 450 participants from Split, Osijek and Zagreb County. Based on the completed standardized questionnaires the target groups of kindergarten children will be classified according to their nutritional status:

1. children who have a developed food allergy
2. children at risk of developing mild, moderate or severe allergic reaction to food
3. children with an allergological indication

The children with allergological indication (c) will be sent for further specialist evaluation, diagonstics and nutritionist advice at CHS.

The investigators will monitor how many kindergarten children have developed food allergy, food intolerance and another allergy (eg. inhalation allergy). Children with another type of allergy will be the refference control.

ELIGIBILITY:
Inclusion Criteria:

* Parental approval
* Children from 1 to 6 years old

Exclusion Criteria:

* Chromosomal abberations
* Neurological disorders that affect oral motorics
* Chronic gastrointestinal disorders
* Severe metabolic disorders

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will include a minimum of 450 preeschool children, aged 1-6 years, from Osijek, Split and Zagreb County.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Development of an IT platform for the introduction of personalized balanced nutrition in kindergartens | 33 months
  IT platform will enable electronic creation and distribution of daily menus, daily collection of information about the food consumed, collecting relevant data and sending nutrition guidelines and instructions to kindergartens and parents.In addition to the above, the system will enable data collection of anthropometric measurements and monitoring of physical activity and send feedback to parents about measurement results. The mentioned system will, among other things, establish a communication link between the Children's Hospital Srebrnjak and kindergartens, which will enhance the exchange of data in real time and the possibility of timely adjustment of the menu.

SECONDARY OUTCOMES:
Differentiation between children with allergies from chlidren's intolerance to food and development of a Register of Allergies | 33 months
  The development of the Register of Allergies will provide pediatricians, general practitioners and specialists with personalized patient information which will ensure the application of appropriate health treatment and gudelines for identifying risk measures and allergic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Srebrnjak, Zagreb, Croatia